CLINICAL TRIAL: NCT04696471
Title: Elucidating Neural Mechanisms of Hypo/Mania Using Theta Burst Stimulation
Brief Title: Effects of Theta Burst Stimulation on the Brain, Behavior, and Clinical Symptoms in Adults With Bipolar Disorder
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mary Phillips, MD MD (Cantab) (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Sponsor-Investigator, Mary Phillips, MD MD (Cantab), Professor, University of Pittsburgh
Organization: University of Pittsburgh (Other)
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: STUDY20060322; R01MH122990 (NIH)
Record Dates: First submitted 2020-12-18; First posted 2021-01-06 (Actual); Last update posted 2026-01-20 (Actual); Status verified 2025-12

CONDITIONS: Bipolar Disorder
Keywords: Bipolar Disorder; Magnetic Resonance Imaging; Transcranial Magnetic Stimulation
MeSH Terms: conditions — Bipolar Disorder | interventions — Transcranial Magnetic Stimulation

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (6):
- Left ventrolateral prefrontal cortex (vlPFC)/Left SS/Left vlPFC sham (Experimental): A random number sequence will be generated for randomization of the 3 cTBS scan session order to which each participant is assigned:
  * left vlPFC cTBS (cTBS applied to the left ventrolateral prefrontal cortex)
  * left SS cTBS (cTBS applied to the left somatosensory area)
  * left vlPFC sham TBS (go through the motions of applying cTBS to the left ventrolateral prefrontal cortex but very low current is administered so that the participant feels like cTBS is being administered even though the current is too low to stimulate brain cells) Participants will know that one session will be a sham, but they will be blinded to which session is the sham.
  Interventions: Device: Continuous Theta Burst Stimulation (cTBS); Device: Sham Continuous Theta Burst Stimulation (Sham cTBS)
- Left vlPFC/Left vlPFC sham/Left SS (Experimental): A random number sequence will be generated for randomization of the 3 cTBS scan session order to which each participant is assigned:
  * left vlPFC cTBS (cTBS applied to the left ventrolateral prefrontal cortex)
  * left SS cTBS (cTBS applied to the left somatosensory area)
  * left vlPFC sham TBS (go through the motions of applying cTBS to the left ventrolateral prefrontal cortex but very low current is administered so that the participant feels like cTBS is being administered even though the current is too low to stimulate brain cells) Participants will know that one session will be a sham, but they will be blinded to which session is the sham.
  Interventions: Device: Continuous Theta Burst Stimulation (cTBS); Device: Sham Continuous Theta Burst Stimulation (Sham cTBS)
- Left SS/Left vlPFC sham/Left vlPFC (Experimental): A random number sequence will be generated for randomization of the 3 cTBS scan session order to which each participant is assigned:
  * left vlPFC cTBS (cTBS applied to the left ventrolateral prefrontal cortex)
  * left SS cTBS (cTBS applied to the left somatosensory area)
  * left vlPFC sham TBS (go through the motions of applying cTBS to the left ventrolateral prefrontal cortex but very low current is administered so that the participant feels like cTBS is being administered even though the current is too low to stimulate brain cells) Participants will know that one session will be a sham, but they will be blinded to which session is the sham.
  Interventions: Device: Continuous Theta Burst Stimulation (cTBS); Device: Sham Continuous Theta Burst Stimulation (Sham cTBS)
- Left SS/Left vlPFC/Left vlPFC sham (Experimental): A random number sequence will be generated for randomization of the 3 cTBS scan session order to which each participant is assigned:
  * left vlPFC cTBS (cTBS applied to the left ventrolateral prefrontal cortex)
  * left SS cTBS (cTBS applied to the left somatosensory area)
  * left vlPFC sham TBS (go through the motions of applying cTBS to the left ventrolateral prefrontal cortex but very low current is administered so that the participant feels like cTBS is being administered even though the current is too low to stimulate brain cells) Participants will know that one session will be a sham, but they will be blinded to which session is the sham.
  Interventions: Device: Continuous Theta Burst Stimulation (cTBS); Device: Sham Continuous Theta Burst Stimulation (Sham cTBS)
- Left vlPFC sham/Left SS/Left vlPFC (Experimental): A random number sequence will be generated for randomization of the 3 cTBS scan session order to which each participant is assigned:
  * left vlPFC cTBS (cTBS applied to the left ventrolateral prefrontal cortex)
  * left SS cTBS (cTBS applied to the left somatosensory area)
  * left vlPFC sham TBS (go through the motions of applying cTBS to the left ventrolateral prefrontal cortex but very low current is administered so that the participant feels like cTBS is being administered even though the current is too low to stimulate brain cells) Participants will know that one session will be a sham, but they will be blinded to which session is the sham.
  Interventions: Device: Continuous Theta Burst Stimulation (cTBS); Device: Sham Continuous Theta Burst Stimulation (Sham cTBS)
- Left vlPFC sham/Left vlPFC/Left SS (Experimental): A random number sequence will be generated for randomization of the 3 cTBS scan session order to which each participant is assigned:
  * left vlPFC cTBS (cTBS applied to the left ventrolateral prefrontal cortex)
  * left SS cTBS (cTBS applied to the left somatosensory area)
  * left vlPFC sham TBS (go through the motions of applying cTBS to the left ventrolateral prefrontal cortex but very low current is administered so that the participant feels like cTBS is being administered even though the current is too low to stimulate brain cells) Participants will know that one session will be a sham, but they will be blinded to which session is the sham.
  Interventions: Device: Continuous Theta Burst Stimulation (cTBS); Device: Sham Continuous Theta Burst Stimulation (Sham cTBS)

INTERVENTIONS:
Device: Continuous Theta Burst Stimulation (cTBS) — cTBS is a brief stimulation of a part of the brain with a magnetic field that passes through the scalp and skull safely. It is FDA-approved as a treatment for psychological conditions including depression; however, this device is not approved for the treatment of adults with Bipolar Disorder I or for use in healthy adults. This research study is using the cTBS off label in all participants (those with and without Bipolar Disorder I) to examine research questions
  Other Names: Transcranial Magnetic Stimulation (TMS)
Device: Sham Continuous Theta Burst Stimulation (Sham cTBS) — Sham cTBS goes through the motions of applying cTBS to the brain but administers very low current so that the participant feels like cTBS is being administered even though the current is too low to stimulate brain cells. Participants will know that one session will be a sham, but they will be blinded to which session is the sham
  Other Names: Sham Transcranial Magnetic Stimulation (Sham TMS)

SUMMARY:
Bipolar Disorder (BD) is a common and highly debilitating psychiatric disorder, however, the predisposing brain mechanisms are poorly understood. Here, the investigators aim to examine the immediate effect of transcranial brain stimulation (TBS) on brain activity and emotions in adults with and without BD as a first stage toward understanding the predisposing brain mechanisms of BD. The investigators hypothesize that TBS will reduce brain activity while playing a game with rewards in all adults, but the TBS will reduce brain activity more in the adults with BD compared to adults without BD. Furthermore, the investigators hypothesize that this reduced brain activity will be associated with reduced BD symptoms, such as negative emotions.

DETAILED DESCRIPTION:
This study aims to examine the effects of noninvasive stimulation on brain activity as measured by functional magnetic resonance imaging (fMRI) in participants with and without Bipolar I Disorder. Eligible participants will undergo 5 study visits: a screening visit, a baseline MRI visit, and 3 cTBS visits. Participants will receive brain stimulation and undergo fMRI scanning at each of the 3 cTBS study visits, however, at one of the visits, the brain stimulation will be a sham. The research associates and participants will be blinded to when the sham occurs, which will be randomized beforehand. Certain information is withheld to protect the scientific integrity of the study design

ELIGIBILITY:
Inclusion Criteria:

1. All participants

   * 18-35 years of age
   * Scoring less than or equal to 8 on the Hamilton Rating Scale for Depression (HRSD) at screen visit
2. Participants with Bipolar Disorder (BD)

   * Diagnosis of Bipolar Disorder I/II (BDI/II) (DSM-5 criteria) in remission (euthymic for >2 months) or with mild-moderate hypomania
   * <15 on the Young Mania Rating Scale
   * Not psychotic
   * <3 on delusions, hallucinations, unusual thought content, and conceptual disorganization items of the Positive and Negative Syndrome Scale (PANSS)
   * Unmedicated or on any combination (except antidepressant monotherapy) of anxiolytics (benzodiazepines, buspirone, pregabalin, hydroxyzine) as needed, and/or atypical antipsychotics, and/or lithium, and/or other mood stabilizers, and/or non-SNRI antidepressants and/or non benzodiazepine hypnotics taken for >2 months, as these are commonly-prescribed medications for BD
3. Participants without Bipolar Disorder

   * No present or lifetime history of BD or psychiatric disorder other than anxiety or non BD mood disorders
   * Not in a current depressive episode
   * No family history of BD

Exclusion Criteria:

1. All participants

   * History of head injury, neurological, pervasive developmental disorder (e.g. autism), systemic medical disease and treatment (medical records, participant report)
   * Family history of epilepsy (TBS exclusion criterion)
   * Use of substances with seizure risk (e.g., stimulants) in the past month, assessed as at screening, baseline, and before each fMRI-cTBS-fMRI session
   * Mini-Mental State Examination score (cognitive state) <24
   * Premorbid National Adult Reading Test Intelligent Quotient estimate<85
   * Visual disturbance: <20/40 Snellen visual acuity
   * Left/mixed handedness
   * History of alcohol/substance use disorder (SUD; all substances, including nicotine), and/or illicit substance use (except cannabis) over the last 6 months (SCID-5). Note: lifetime/present cannabis use (at non-abuse (<3 times in the past month) and non SUD levels) will be allowed, given its common usage in BD and young adults. Cannabis SUD over the last 6 months will not be allowed. Urine tests on scan days will exclude current illicit substance use (except cannabis). Salivary alcohol tests on scan days will exclude intoxicated individuals
   * Binge drinking in the week before, and/or >3 units/day for the 3 days before, and/or alcohol in the last 12 hrs before, any cTBS scan day, confirmed at screening and scan days (to avoid TBS during alcohol withdrawal). Alcohol/nicotine/ caffeine/cannabis use (below SCID-5 SUD, binge levels) will be allowed, and used as covariates
   * MRI exclusion criteria: metallic objects, e.g., surgical implants; claustrophobia; proneness; positive pregnancy test for females (performed at the MRRC) or self-report pregnancy
   * Inability to understand English
   * <18 years of age or >35 year of age

     * SNRI antidepressants and bupropion will not be allowed, as they can elevate seizure risk, a contraindication for TBS
     * Scoring greater than or equal to 8 on HRSD and in depressive episode is confirmed on SCID-5 at screen visit
     * Scoring greater than or equal to 18 on HRSD at any visit
     * In current depressive episode
2. Participants with Bipolar Disorder

   * BD diagnosis other than BDI/II
   * More severe hypo/mania (YMRS>15)
   * Psychosis
   * Using psychotropic medications other than those allowed in inclusion criteria
3. Participants without Bipolar Disorder

   * Present/ lifetime history of any psychiatric disorder other than anxiety and non BD mood disorders
   * Family history of of BD

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 146 (Actual)
Dates: Start 2021-04-06 (Actual); Primary Completion 2025-10-24 (Actual); Study Completion 2025-10-24 (Actual)

PRIMARY OUTCOMES:
Reward expectancy-related left ventrolateral prefrontal cortex activity | Change in magnitude immediately before and immediately after each cTBS condition at scan visits (30-60 mins)
  The difference in magnitude between pre and post cTBS scans for each cTBS condition of the extracted blood oxygen level-dependent (BOLD) signal from the left ventrolateral prefrontal cortex to the uncertain reward expectancy regressor during performance of the reward task
Reward expectancy-related right ventrolateral prefrontal cortex activity | Change in magnitude immediately before and immediately after each cTBS condition at scan visits (30-60 mins)
  The difference in magnitude between pre and post cTBS scans for each cTBS condition of the extracted BOLD signal from the right ventrolateral prefrontal cortex to the uncertain reward expectancy regressor during performance of the reward task
Reward expectancy-related left ventral striatum activity | Change in magnitude immediately before and immediately after each cTBS condition at scan visits (30-60 mins)
  The difference in magnitude between pre and post cTBS scans for each cTBS condition of the extracted BOLD signal from the left ventral striatum to the uncertain reward expectancy regressor during performance of the reward task
Reward expectancy-related right ventral striatum activity | Change in magnitude immediately before and immediately after each cTBS condition at scan visits (30-60 mins)
  The difference in magnitude between pre and post cTBS scans for each cTBS condition of the extracted BOLD signal from the left ventral striatum to the uncertain reward expectancy regressor during performance of the reward task
Reward expectancy-related left orbitofrontal cortex activity | Change in magnitude immediately before and immediately after each cTBS condition at scan visits (30-60 mins)
  The difference in magnitude between pre and post cTBS scans for each cTBS condition of the extracted BOLD signal from the left orbitofrontal cortex to the uncertain reward expectancy regressor during performance of the reward task
Reward expectancy-related right orbitofrontal cortex activity | Change in magnitude immediately before and immediately after each cTBS condition at scan visits (30-60 mins)
  The difference in magnitude between pre and post cTBS scans for each cTBS condition of the extracted BOLD signal from the left orbitofrontal cortex to the uncertain reward expectancy regressor during performance of the reward task
Reward expectancy-related midline rostral anterior cingulate cortex (rACC) activity | Change in magnitude immediately before and immediately after each cTBS condition at scan visits (30-60 mins)
  The difference in magnitude between pre and post cTBS scans for each cTBS condition of the extracted BOLD signal from the midline rostral anterior cingulate cortex (rACC) to the uncertain reward expectancy regressor during performance of the reward task
Reward expectancy-related midline dorsal anterior cingulate cortex activity | Change in magnitude immediately before and immediately after each cTBS condition at scan visits (30-60 mins)
  The difference in magnitude between pre and post cTBS scans for each cTBS condition of the extracted BOLD signal from the midline dorsal anterior cingulate cortex to the uncertain reward expectancy regressor during performance of the reward task
Reward expectancy-related left amygdala activity | Change in magnitude immediately before and immediately after each cTBS condition at scan visits (30-60 mins)
  The difference in magnitude between pre and post cTBS scans for each cTBS condition of the extracted BOLD signal from the left amygdala to the uncertain reward expectancy regressor during performance of the reward task
Reward expectancy-related right amygdala activity | Change in magnitude immediately before and immediately after each cTBS condition at scan visits (30-60 mins)
  The difference in magnitude between pre and post cTBS scans for each cTBS condition of the extracted BOLD signal from the left amygdala to the uncertain reward expectancy regressor during performance of the reward task
Reward expectancy-related left ventrolateral prefrontal cortex-right ventrolateral prefrontal cortex functional connectivity | Change in magnitude immediately before and immediately after each cTBS condition at scan visits (30-60 mins)
  The difference in magnitude between pre and post cTBS scans for each cTBS condition of the extracted parameter estimate for functional connectivity between the left and right ventrolateral prefrontal cortices to the uncertain reward expectancy regressor during performance of the reward task
Reward expectancy-related left ventrolateral prefrontal cortex-left ventral striatum functional connectivity | Change in magnitude immediately before and immediately after each cTBS condition at scan visits (30-60 mins)
  The difference in magnitude between pre and post cTBS scans for each cTBS condition of the extracted parameter estimate for functional connectivity between the left ventrolateral prefrontal cortex and left ventral striatum to the uncertain reward expectancy regressor during performance of the reward task
Reward expectancy-related left ventrolateral prefrontal cortex-right ventral striatum functional connectivity | Change in magnitude immediately before and immediately after each cTBS condition at scan visits (30-60 mins)
  The difference in magnitude between pre and post cTBS scans for each cTBS condition of the extracted parameter estimate for functional connectivity between the left ventrolateral prefrontal cortex and right ventral striatum to the uncertain reward expectancy regressor during performance of the reward task
Reward expectancy-related left ventrolateral prefrontal cortex-left orbitofrontal cortex functional connectivity | Change in magnitude immediately before and immediately after each cTBS condition at scan visits (30-60 mins)
  The difference in magnitude between pre and post cTBS scans for each cTBS condition of the extracted parameter estimate for functional connectivity between the left ventrolateral prefrontal cortex and left orbitofrontal cortex to the uncertain reward expectancy regressor during performance of the reward task
Reward expectancy-related left ventrolateral prefrontal cortex-right orbitofrontal cortex functional connectivity | Change in magnitude immediately before and immediately after each cTBS condition at scan visits (30-60 mins)
  The difference in magnitude between pre and post cTBS scans for each cTBS condition of the extracted parameter estimate for functional connectivity between the left ventrolateral prefrontal cortex and right orbitofrontal cortex to the uncertain reward expectancy regressor during performance of the reward task
Reward expectancy-related left ventrolateral prefrontal cortex-midline rostral anterior cingulate cortex functional connectivity | Change in magnitude immediately before and immediately after each cTBS condition at scan visits (30-60 mins)
  The difference in magnitude between pre and post cTBS scans for each cTBS condition of the extracted parameter estimate for functional connectivity between the left ventrolateral prefrontal cortex and midline rACC to the uncertain reward expectancy regressor during performance of the reward task
Reward expectancy-related left ventrolateral prefrontal cortex-midline dorsal anterior cingulate cortex functional connectivity | Change in magnitude immediately before and immediately after each cTBS condition at scan visits (30-60 mins)
  The difference in magnitude between pre and post cTBS scans for each cTBS condition of the extracted parameter estimate for functional connectivity between the left ventrolateral prefrontal cortex and midline dorsal anterior cingulate cortex to the uncertain reward expectancy regressor during performance of the reward task
Reward expectancy-related left ventrolateral prefrontal cortex-left amygdala functional connectivity | Change in magnitude immediately before and immediately after each cTBS condition at scan visits (30-60 mins)
  The difference in magnitude between pre and post cTBS scans for each cTBS condition of the extracted parameter estimate for functional connectivity between the left ventrolateral prefrontal cortex and left amygdala to the uncertain reward expectancy regressor during performance of the reward task
Reward expectancy-related left ventrolateral prefrontal cortex-right amygdala functional connectivity | Change in magnitude immediately before and immediately after each cTBS condition at scan visits (30-60 mins)
  The difference in magnitude between pre and post cTBS scans for each cTBS condition of the extracted parameter estimate for functional connectivity between the left ventrolateral prefrontal cortex and right amygdala to the uncertain reward expectancy regressor during performance of the reward task

SECONDARY OUTCOMES:
Reward expectancy-related left ventrolateral prefrontal cortex wholebrain functional connectivity | Change in magnitude immediately before and immediately after each cTBS condition at scan visits (30-60 mins)
  The difference in magnitude between pre and post cTBS for each cTBS condition of the extracted parameter estimate for functional connectivity between the left ventrolateral prefrontal cortex and the whole brain to the uncertain reward expectancy regressor during performance of the reward task
Left ventrolateral prefrontal cortex activity | Change in magnitude immediately before and immediately after each cTBS condition at scan visits (30-60 mins)
  The difference in magnitude between pre and post cTBS scans for each cTBS condition of the extracted BOLD signal in the left ventrolateral prefrontal cortex to the contrast of possible win vs. neutral control conditions
Right ventrolateral prefrontal cortex activity | Change in magnitude immediately before and immediately after each cTBS condition at scan visits (30-60 mins)
  The difference in magnitude between pre and post cTBS scans for each cTBS condition of the extracted BOLD signal in the right ventrolateral prefrontal cortex to the contrast of possible win vs. neutral control conditions
Left ventral striatum activity | Change in magnitude immediately before and immediately after each cTBS condition at scan visits (30-60 mins)
  The difference in magnitude between pre and post cTBS scans for each cTBS condition of the extracted BOLD signal in the left ventral striatum to the contrast of possible win vs. neutral control conditions
Right ventral striatum activity | Change in magnitude immediately before and immediately after each cTBS condition at scan visits (30-60 mins)
  The difference in magnitude between pre and post cTBS scans for each cTBS condition of the extracted BOLD signal in the right ventral striatum to the contrast of possible win vs. neutral control conditions
Left orbitofrontal cortex activity | Change in magnitude immediately before and immediately after each cTBS condition at scan visits (30-60 mins)
  The difference in magnitude between pre and post cTBS scans for each cTBS condition of the extracted BOLD signal in the left orbitofrontal cortex to the contrast of possible win vs. neutral control conditions
Right orbitofrontal cortex activity | Change in magnitude immediately before and immediately after each cTBS condition at scan visits (30-60 mins)
  The difference in magnitude between pre and post cTBS scans for each cTBS condition of the extracted BOLD signal in the right orbitofrontal cortex to the contrast of possible win vs. neutral control conditions
Midline rostral anterior cingulate cortex activity | Change in magnitude immediately before and immediately after each cTBS condition at scan visits (30-60 mins)
  The difference in magnitude between pre and post cTBS scans for each cTBS condition of the extracted BOLD signal in the midline rostral anterior cingulate cortex to the contrast of possible win vs. neutral control conditions
Midline dorsal anterior cingulate cortex activity | Change in magnitude immediately before and immediately after each cTBS condition at scan visits (30-60 mins)
  The difference in magnitude between pre and post cTBS scans for each cTBS condition of the extracted BOLD signal in the midline dorsal anterior cingulate cortex to the contrast of possible win vs. neutral control conditions
Left amygdala activity | Change in magnitude immediately before and immediately after each cTBS condition at scan visits (30-60 mins)
  The difference in magnitude between pre and post cTBS scans for each cTBS condition of the extracted BOLD signal in the left amygdala to the contrast of possible win vs. neutral control conditions
Right amygdala activity | Change in magnitude immediately before and immediately after each cTBS condition at scan visits (30-60 mins)
  The difference in magnitude between pre and post cTBS scans for each cTBS condition of the extracted BOLD signal in the right amygdala to the contrast of possible win vs. neutral control conditions
Left ventral lateral prefrontal cortex-wholebrain functional connectivity | Change in magnitude immediately before and immediately after each cTBS condition at scan visits (30-60 mins)
  The difference in magnitude between pre and post cTBS scans for each cTBS condition of the extracted parameter estimates of functional connectivity between the left ventrolateral prefrontal cortex and the wholebrain to the contrast of possible win vs. neutral control conditions
Prediction error-related left ventral striatum activity | Change in magnitude immediately before and immediately after each cTBS condition at scan visits (30-60 mins)
  The difference in magnitude between pre and post cTBS scans for each cTBS condition of the extracted BOLD signal in the left ventral striatum to the prediction error regressor
Prediction error-related right ventral striatum activity | Change in magnitude immediately before and immediately after each cTBS condition at scan visits (30-60 mins)
  The difference in magnitude between pre and post cTBS scans for each cTBS condition of the extracted BOLD signal in the right ventral striatum to the prediction error regressor
Prediction error-related left ventral striatum-wholebrain functional connectivity | Change in magnitude immediately before and immediately after each cTBS condition at scan visits (30-60 mins)
  The difference in magnitude between pre and post cTBS scans for each cTBS condition of the extracted parameter estimates of resting state functional connectivity between the left ventral striatum and the wholebrian to the prediction error regressor
Prediction error-related right ventral striatum-wholebrain functional connectivity | Change in magnitude immediately before and immediately after each cTBS condition at scan visits (30-60 mins)
  The difference in magnitude between pre and post cTBS scans for each cTBS condition of the extracted parameter estimates of resting state functional connectivity between the right ventral striatum and the wholebrain

OTHER OUTCOMES:
Left ventrolateral prefrontal cortex-wholebrain resting state functional connectivity | Change in magnitude immediately before and immediately after each cTBS condition at scan visits (30-60 mins)
  The difference in magnitude between pre and post cTBS scans for each cTBS condition of the extracted parameter estimates of resting state functional connectivity between the left ventrolateral prefrontal cortex and the wholebrain
Left ventrolateral prefrontal cortex-right ventrolateral prefrontal cortex resting state functional connectivity | Change in magnitude immediately before and immediately after each cTBS condition at scan visits (30-60 mins)
  The difference in magnitude between pre and post cTBS scans for each cTBS condition of the extracted parameter estimates of resting state functional connectivity between the left and right ventrolateral prefrontal cortices
Left ventrolateral prefrontal cortex-left ventral striatum resting state functional connectivity | Change in magnitude immediately before and immediately after each cTBS condition at scan visits (30-60 mins)
  The difference in magnitude between pre and post cTBS scans for each cTBS condition of the extracted parameter estimates of resting state functional connectivity between the left ventrolateral prefrontal cortex and the left ventral striatum
Left ventrolateral prefrontal cortex-right ventral striatum resting state functional connectivity | Change in magnitude immediately before and immediately after each cTBS condition at scan visits (30-60 mins)
  The difference in magnitude between pre and post cTBS scans for each cTBS condition of the extracted parameter estimates of resting state functional connectivity between the left ventrolateral prefrontal cortex and the right ventral striatum
Left ventrolateral prefrontal cortex-left orbitofrontal cortex resting state functional connectivity | Change in magnitude immediately before and immediately after each cTBS condition at scan visits (30-60 mins)
  The difference in magnitude between pre and post cTBS scans for each cTBS condition of the extracted parameter estimates of resting state functional connectivity between the left ventrolateral prefrontal cortex and the left orbitofrontal cortex
Left ventrolateral prefrontal cortex-right orbitofrontal cortex resting state functional connectivity | Change in magnitude immediately before and immediately after each cTBS condition at scan visits (30-60 mins)
  The difference in magnitude between pre and post cTBS scans for each cTBS condition of the extracted parameter estimates of resting state functional connectivity between the left ventrolateral prefrontal cortex and the right orbitofrontal cortex
Left ventrolateral prefrontal cortex-midline rostral anterior cingulate cortex resting state functional connectivity | Change in magnitude immediately before and immediately after each cTBS condition at scan visits (30-60 mins)
  The difference in magnitude between pre and post cTBS scans for each cTBS condition of the extracted parameter estimates of resting state functional connectivity between the left ventrolateral prefrontal cortex and the midline rostral anterior cingulate cortex
Left ventrolateral prefrontal cortex-midline dorsal anterior cingulate cortex resting state functional connectivity | Change in magnitude immediately before and immediately after each cTBS condition at scan visits (30-60 mins)
  The difference in magnitude between pre and post cTBS scans for each cTBS condition of the extracted parameter estimates of resting state functional connectivity between the left ventrolateral prefrontal cortex and the midline dorsal anterior cingulate cortex
Left ventrolateral prefrontal cortex-left amygdala resting state functional connectivity | Change in magnitude immediately before and immediately after each cTBS condition at scan visits (30-60 mins)
  The difference in magnitude between pre and post cTBS scans for each cTBS condition of the extracted parameter estimates of resting state functional connectivity between the left ventrolateral prefrontal cortex and the left amygdala
Left ventrolateral prefrontal cortex-right amygdala resting state functional connectivity | Change in magnitude immediately before and immediately after each cTBS condition at scan visits (30-60 mins)
  The difference in magnitude between pre and post cTBS scans for each cTBS condition of the extracted parameter estimates of resting state functional connectivity between the left ventrolateral prefrontal cortex and the right amygdala

CONTACTS AND LOCATIONS:
Overall Officials: Mary Phillips, MD, MD, Principal Investigator — University of Pittsburgh; Fabio Ferrarelli, MD, PhD, Principal Investigator — University of Pittsburgh
Locations (1):
- University of Pittsburgh, Pittsburgh, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: Yes
The investigators will complete and submit a National Data Archive (NDA) Data Sharing Agreement within 6 months of the Notice of Award Issue date. Study staff will upload data dictionary to the NDA website, and will review the NDA data definition for the measures collected and define the project's data definition harmonized to that standard. For measures not yet defined, project staff will work with the NDA staff to define the measure following NDA best practices. Informed consent will be collected from study participants that allows for broad sharing of participants' de-identified data. Study staff will use participants' personally identifiable information to generate NDA Global Unique Identifier (GUID) numbers for study participants.
  All data will be identified by GUID numbers only prior to submission to the NDA database. Data transfer procedures will be in accordance with all Institutional Review Board guidelines and federal regulations including HIPAA.
Time Frame: Raw data and data from descriptive/raw measures will be submitted on a semi-annual basis by July 15 and January 15 or the next business day. We also agree to submit to NDA the analyzed data yielded in our project (i.e., 12 months after accomplishment of each primary aim or objective, or immediately upon publication of the project's primary results, whichever occurs first). The PIs reserve the right to publish on the stated aims in a timely manner during the period of the award. Data will be available for addressing other research questions (i.e. which are not described in funded/pending grants) as soon as the data have been checked for accuracy (a period which will be no later than one year after the completion of each assessment). After the award has ended, the study investigators will continue to test the stated aims, but will also continue to solicit collaborations with outside researchers and to consider data requests in a timely manner.
Access Criteria: Outside investigators must submit a 1)proposal of the study aims, hypotheses, variables/constructs, analytic approach, and estimated duration of the proposed research; 2)resume, qualifications, source of financial support, and conflict of interest statement; 3)sign a data-sharing agreement and confidentiality statement that stipulates using the data for the stated research purposes only, securing the data using appropriate computer technology, not manipulating the data in order to identify participants, acknowledging the grant that supported data collection and management in publications/presentations, and destroying or returning the data after analyses are complete; 4)obtain approval from their Institutional Review Board, and along with other staff members who have access to the data, submit certificates of the University of Pittsburgh Education and Certification Program in Research Practice Fundamentals or provide written documentation pf similar human subjects protection training.

DOCUMENTS (1):
  • Informed Consent Form (2025-05-13): https://cdn.clinicaltrials.gov/large-docs/71/NCT04696471/ICF_000.pdf